CLINICAL TRIAL: NCT03196362
Title: Impacts of Sequential Treatment Using Fixed Dose Pioglitazone/Metformin Combination Following Short-term Intensive Insulin Treatment on Long-term Blood Glucose Control and β-Cell Function in Patients With Newly Diagnosed Type 2 Diabetes
Brief Title: Impacts of PIO/MET Following Short-term Intensive Insulin Treatment in Newly Diagnosed Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanbing Li, Director of Endocrinology and Metabolism Department, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20160145
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: short-term intensive insulin therapy; pioglitazone; metformin; remission; sequential therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIO/MET (Active Comparator): one fixed dose pioglitazone/metformin (15mg/500mg) tablet will be orally administrated twice daily
  Interventions: Drug: Pioglitazone + Metformin
- placebo (Placebo Comparator): one tablet of placebo will be given twice daily
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Pioglitazone + Metformin — One tablet of fixed dose of Pioglitazone/ Metformin (15mg/30mg) will be given twice daily
  Arms: PIO/MET
Drug: Placebo Oral Tablet — One tablet of placebo will be given twice daily
  Arms: placebo

SUMMARY:
Short-term intensive insulin therapy (SIIT) induces glycemic remission in patients with newly diagnosed type 2 diabetes. But remission rate reduces over time. This study aims to investigate whether sequential treatments using fixed dose combination of pioglitazone/metformin (15mg/500mg) after SIIT can improve clinical outcomes inpatients with newly diagnosed type 2 diabetes.

We plan to include 50 patients with newly diagnosed type 2 diabetes who are drug naïve and meet the inclusive criteria will be enrolled. After baseline assessments, SIIT will be applied to all patients using insulin pump to achieve and maintain euglycemia for 2 weeks. After completion of intensive treatment, insulin pump will be stopped. Patients were randomly assigned into either of the following two groups: PIO/MET group: pioglitazone/metformin (15mg/500mg) will be orally administrated twice daily to the subjects for 12 weeks; placebo group: placebo is given twice daily to all subjects for 12 weeks. Afterwards, patients will be followed up for 48 weeks. Primary endpoint is difference in remission rate at the end of study. Secondary endpoints include proportion of patients who achieve glycosylated hemoglobin A1C <7% at the end of study; differences in β-cell function , insulin sensitivity and incidence of adverse events among treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed type 2 diabetes who have never received any hypoglycemic treatment;
2. Fasting plasma glucose (FPG) between 7.0 mmol/l (126 mg/dl) and 16.7 mmol/l (300 mg/dl); glycosylated hemoglobin A1C>8.5%;
3. Aged between 25 and 65 years,
4. Body mass index (BMI) 22-35 kg/m2.

Exclusion Criteria:

1. Type 1 diabetes or special type of diabetes;
2. Acute diabetic complications of diabetes (DKA, HHS and lactic acidosis etc.)
3. Serious microvascular complications: proliferative stage of retinopathy; urine AER >300 mg/g or urine protein positive, quantification >0.5 g/d; uncontrolled painful diabetic neuropathy and significant diabetic autonomic neuropathy;
4. Severe macrovascular complications: acute cerebrovascular accident, acute coronary syndrome, vascular intervention for peripheral arterial disease or amputation requiring hospitalization within 12 months prior to enrollment;
5. Persistently increased blood pressure >180/110 mmHg;
6. Blood creatinine clearance less than 50 ml/min, alanine aminotransferase ≥2.5×upper limit of normal, total bilirubin ≥1.5×upper limit of normal;
7. Hemoglobin <100 g/L or need regular blood transfusion;
8. Use of drugs that may influence blood glucose within 12 weeks;
9. Systemic infection or serious concomitant disease; patients with malignancy or chronic diarrhea;
10. Uncontrolled endocrine gland dysfunction;
11. Patients with mental or communication disorders;
12. Chronic cardiac insufficiency, heart function class III and above;
13. Pregnant women, lactating women and women of child bearing age who are not willing to take contraception during the study;
14. Subjects who don't cooperate, cannot be followed up or have difficulty in completing the study considered by the investigator.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Remission rate | 48 weeks
  Remission rate at the end of the study in each group

SECONDARY OUTCOMES:
β-cell function | 48 weeks
  Difference in β-cell secretion capacity at the end of follow up between treatment groups
Insulin sensitivity | 48 weeks
  Difference in insulin sensitivity at the end of follow up between treatment groups
glycemic control | 48 weeks
  proportion of patients who achieve A1C<7% at the end of follow-up
Adverse events | 48 weeks
  difference in AEs at the end of follow-up between treatment groups

CONTACTS AND LOCATIONS:
Locations (1):
- endocrinology department of the first affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No